CLINICAL TRIAL: NCT02162355
Title: Randomized, Double-blind, Placebo-controlled Study for the Assessment of Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics, of Multiple Oral Doses of GLPG0634 in Japanese and Caucasian Healthy Subjects
Brief Title: Multiple Ascending Dose Study of GLPG0634 in Japanese and Caucasian Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GLPG0634-CL-110; 2013-004408-21 (EudraCT Number)
Record Dates: First submitted 2014-06-11; First posted 2014-06-12 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG0634; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GLPG0634 in Japanese subjects (Experimental): Per panel, 6 Japanese healthy subjects will receive one of the three doses (50 mg, 100 mg or 200 mg) of GLPG0634 as tablets once daily for 10 days
  Interventions: Drug: GLPG0634 50 mg; Drug: GLPG0634 100 mg; Drug: GLPG0634 200 mg
- Placebo in Japanese healthy subjects (Placebo Comparator): Per panel, 2 or 4 (last panel only) Japanese healthy subjects will receive placebo as tablets once daily for 10 days
  Interventions: Drug: Placebo
- GLPG0634 in Caucasian subjects (Experimental): In the last panel, 6 Caucasian healthy subjects will receive one dose of GLPG0634 (200 mg) as tablets once daily for 10 days
  Interventions: Drug: GLPG0634 200 mg
- Placebo in Caucasian healthy subjects (Placebo Comparator): In the last panel, 4 Caucasian healthy subjects will receive receive placebo as tablets once daily for 10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG0634 50 mg — 2 tablets of 25 mg GLPG0634 once daily for 10 days
  Other Names: 50 mg GLPG0634 as tablets
  Arms: GLPG0634 in Japanese subjects
Drug: GLPG0634 100 mg — 1 tablet of 100 mg GLPG0634 once daily for 10 days
  Other Names: 100 mg GLPG0634 as tablets
  Arms: GLPG0634 in Japanese subjects
Drug: GLPG0634 200 mg — 2 tablets of 100 mg GLPG0634 once daily for 10 days
  Other Names: 200 mg GLPG0634 as tablets
  Arms: GLPG0634 in Caucasian subjects; GLPG0634 in Japanese subjects
Drug: Placebo — 1 or 2 matching placebo tablets once daily for 10 days
  Other Names: Placebo as matching tablets
  Arms: Placebo in Caucasian healthy subjects; Placebo in Japanese healthy subjects

SUMMARY:
The purpose of this multiple ascending dose study is to characterize the safety, tolerability, and the amount of GLPG0634 present in the blood and urine (pharmacokinetics) of once daily oral administrations of GLPG0634 at 3 different dose levels for 10 days in Japanese healthy subjects.

Furthermore, the study will compare the safety, tolerability, pharmacokinetics, and effects of GLPG0634 on mechanism of action-related parameters in the blood (pharmacodynamics) of once daily oral administrations of GLPG0634 given at one dose level for 10 days in Japanese vs Caucasian healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Japanese or Caucasian subjects between 20-65 years of age (included)
* Subjects must have a body mass index between 18-28 kg/m² (included)
* Subjects must be judged to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram and laboratory profile

Exclusion Criteria:

* A subject with a known hypersensitivity to ingredients of the study drug or a significant allergic reaction to any drug
* Concurrent participation or participation within 3 months prior to the initial study drug administration in a drug/device or biologic investigational research study
* A subject with active drug or alcohol abuse within 2 years prior to the initial study drug administration
* Subject expresses current desire to have (more) children
* Female subject is less than 6 months post-partum, post-abortion or post lactation prior to study drug administration or is pregnant or breastfeeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The number of subjects with adverse events | From screening up to 10 days after last dose (Day 20)
  To evaluate the safety and tolerability of GLPG0634 versus placebo in Japanese subjects at different dose levels, and between Japanese and Caucasian subjects at the highest dose level of GLPG0634 tested in terms of adverse events (AEs)
The number of subjects with abnormal laboratory parameters | From screening up to 10 days after last dose (Day 20)
  To evaluate the safety and tolerability of GLPG0634 versus placebo in Japanese subjects at different dose levels, and between Japanese and Caucasian subjects at the highest dose level of GLPG0634 tested in terms of abnormal laboratory parameters
The number of subjects with abnormal vital signs | From screening up to 10 days after last dose (Day 20)
  To evaluate the safety and tolerability of GLPG0634 versus placebo in Japanese subjects at different dose levels, and between Japanese and Caucasian subjects at the highest dose level of GLPG0634 tested in terms of abnormal vital signs
The number of subjects with abnormal electrocardiogram | From screening up to 10 days after last dose (Day 20)
  To evaluate the safety and tolerability of GLPG0634 versus placebo in Japanese subjects at different dose levels, and between Japanese and Caucasian subjects at the highest dose level of GLPG0634 tested in terms of abnormal electrocardiogram
The number of subjects with abnormal physical examination | From screening up to 10 days after last dose (Day 20)
  To evaluate the safety and tolerability of GLPG0634 versus placebo in Japanese subjects at different dose levels, and between Japanese and Caucasian subjects at the highest dose level of GLPG0634 tested in terms of abnormal physical examination
The amount of GLPG0634 and metabolite in plasma and urine | Between Day 1 before dosing and Day 13 (72 hours after last dose)
  To characterize the amount of GLPG0634 and metabolite in plasma and urine over time - pharmacokinetics (PK) - in Japanese subjects at different dose levels, and between Japanese and Caucasian subjects at the highest dose level of GLPG0634 tested
  Safety Issue?:
  No

SECONDARY OUTCOMES:
The amount of GLPG0634 mechanism-of-action-related biomarkers in blood | Between Day 1 before dosing and Day 11 (24 hours after last dose)
  To characterize the effects of GLPG0634 on mechanism of action-related biomarkers in the blood over time - pharmacodynamics (PD) - in Japanese and Caucasian subjects at the highest dose level of GLPG0634 tested

CONTACTS AND LOCATIONS:
Overall Officials: Pille Harrison, MD, Study Director — Galapagos NV
Locations (1):
- Hammersmith Medicines Research (HMR), London, United Kingdom